CLINICAL TRIAL: NCT03360643
Title: Point-of-Care Ultrasonography for Intussusception: A Randomized Noninferiority Trial
Brief Title: Point-of-Care Ultrasonography for Intussusception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Principal Investigator, Kelly Bergmann, DO, MS, Emergency Research Director, Pediatric Emergency Medicine, Children's Hospitals and Clinics of Minnesota
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1711-153
Record Dates: First submitted 2017-11-20; First posted 2017-12-04 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Intussusception; Emergencies
Keywords: Point-of-care ultrasound; Intussusception; Pediatric Emergency Medicine; Ultrasound
MeSH Terms: conditions — Intussusception; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Point-of-care ultrasound prior to radiology ultrasound (Active Comparator)
  Interventions: Diagnostic Test: Point-of-care ultrasound prior to radiology ultrasound
- Radiology-performed ultrasound (Active Comparator)
  Interventions: Diagnostic Test: Radiology-performed ultrasound

INTERVENTIONS:
Diagnostic Test: Point-of-care ultrasound prior to radiology ultrasound — Point-of-care ultrasound performed by pediatric emergency medicine physicians prior to radiology-performed ultrasound
  Arms: Point-of-care ultrasound prior to radiology ultrasound
Diagnostic Test: Radiology-performed ultrasound — Ultrasound performed an ultrasound technician and/or radiologist, and interpreted by a radiologist
  Arms: Radiology-performed ultrasound

SUMMARY:
Pediatric emergency medicine (PEM) physicians are increasingly utilizing point-of-care ultrasound (POCUS). There is currently limited data regarding POCUS evaluation for intussusception in pediatric patients. To better understand the role of POCUS for identification of intussusception, the investigators plan to conduct a randomized, noninferiority study comparing POCUS and radiology-performed ultrasound (RADUS), utilizing experienced sonographers across multiple institutions.

DETAILED DESCRIPTION:
Intussusception is the most common causes of bowel obstruction among children less than 6 years of age. Limited abdominal ultrasonography is recommended as the initial screening study, prior to enema or surgical reduction for definitive treatment. Although ultrasonography is typically performed by ultrasound technicians and interpreted by radiologists, recently published guidelines include identification of intussusception as an adjunct POCUS application for emergency physicians to use at the bedside.

Two previous studies have investigated POCUS use by PEM physicians for the diagnosis of intussusception, both of which largely incorporated novice sonographers with limited training in bowel ultrasonography. Only one previous prospective investigation has investigated POCUS for the identification of intussusception, with a reported POCUS sensitivity of 85% (95% confidence interval 54-97%) and specificity of 97% (95% confidence interval 89-99%) when compared to RADUS. In contrast, the sensitivity and specificity of RADUS have been reported to range from 98-100% and 88-98%, respectively, when compared to enema or surgical reduction. Given the limited evidence available, it remains unclear whether POCUS performs similar to RADUS in terms of diagnostic accuracy.

The primary aim of this study is to determine whether POCUS is noninferior to RADUS for the detection of intussusception. The secondary aims are to determine whether rates of serious complications or resource utilization measures differ among patients randomly assigned to receive POCUS prior to RADUS or RADUS alone. The investigators hypothesize that diagnostic accuracy, expressed as sensitivity and specificity, is similar for POCUS and RADUS, and that rates of serious complications and resource utilization measures do not differ across groups.

ELIGIBILITY:
Inclusion Criteria:

* Children 3 months through 6 years of age;
* Clinical suspicion for intussusception per treating emergency physician.

Exclusion Criteria:

* Need for critical care resuscitation (intubation or vasopressors);
* Emergent situation where the treating provider determines that POCUS prior to RADUS may interfere with clinical care.

Ages: 3 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 256 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of POCUS and RADUS for clinically important intussusception, expressed as sensitivity and specificity | 2 years from start of enrollment

SECONDARY OUTCOMES:
Rates of recurrent intussusception | 2 years from start of enrollment
  The number of patients with recurrent intussusception in each study arm
Rate of peritonitis | 2 years from start of enrollment
  The number of patients with peritonitis in each study arm
Rate of bowel perforation | 2 years from start of enrollment
  The number of patients with bowel perforation in each study arm
Rate of intestinal obstruction | 2 years from start of enrollment
  The number of patients with intestinal obstruction in each study arm
Rate of shock | 2 years from start of enrollment
  The number of patients with shock in each study arm
Rate of death | 2 years from start of enrollment
  The number of deaths in each study arm
Emergency Department length of stay | 2 years from start of enrollment
Hospital length of stay (for patients admitted to the hospital) | 2 years from start of enrollment
Emergency Department laboratory investigations | 2 years from start of enrollment
  The total number of laboratory investigations obtained per patient
Radiology studies | 2 years after start of enrollment
  The total number of radiology studies obtained per patient
Emergency Department return visit at 3 days | 3 days after the index ED visit
  Return ED visit 3 days after index ED visit
Emergency Department return visit at 7 days | 7 days after the index ED visit
  Return ED visit 7 days after index ED visit
Differentiation of ileocolic and ileoileal intussusception, measured in centimeters | 2 years from start of enrollment
  Ileocolic intussusception will be identified by a maximal cross-sectional diameter of greater than or equal to 2.5 cm; and ileoileal intussusception will be considered less than 2.5 cm in maximal cross-sectional diameter

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Waseem M, Rosenberg HK. Intussusception. Pediatr Emerg Care. 2008 Nov;24(11):793-800. doi: 10.1097/PEC.0b013e31818c2a3e. PMID 19018227
- [Background] Hryhorczuk AL, Strouse PJ. Validation of US as a first-line diagnostic test for assessment of pediatric ileocolic intussusception. Pediatr Radiol. 2009 Oct;39(10):1075-9. doi: 10.1007/s00247-009-1353-z. Epub 2009 Aug 6. PMID 19657636
- [Background] Daneman A, Navarro O. Intussusception. Part 1: a review of diagnostic approaches. Pediatr Radiol. 2003 Feb;33(2):79-85. doi: 10.1007/s00247-002-0832-2. Epub 2002 Nov 19. PMID 12557062
- [Background] Daneman A, Navarro O. Intussusception. Part 2: An update on the evolution of management. Pediatr Radiol. 2004 Feb;34(2):97-108; quiz 187. doi: 10.1007/s00247-003-1082-7. Epub 2003 Nov 21. PMID 14634696
- [Background] American College of Emergency Physicians. Emergency ultrasound guidelines. Ann Emerg Med. 2009 Apr;53(4):550-70. doi: 10.1016/j.annemergmed.2008.12.013. No abstract available. PMID 19303521
- [Background] Vieira RL, Hsu D, Nagler J, Chen L, Gallagher R, Levy JA; American Academy of Pediatrics. Pediatric emergency medicine fellow training in ultrasound: consensus educational guidelines. Acad Emerg Med. 2013 Mar;20(3):300-6. doi: 10.1111/acem.12087. PMID 23517263
- [Background] Lam SH, Wise A, Yenter C. Emergency bedside ultrasound for the diagnosis of pediatric intussusception: a retrospective review. World J Emerg Med. 2014;5(4):255-8. doi: 10.5847/wjem.j.issn.1920-8642.2014.04.002. PMID 25548597
- [Background] Riera A, Hsiao AL, Langhan ML, Goodman TR, Chen L. Diagnosis of intussusception by physician novice sonographers in the emergency department. Ann Emerg Med. 2012 Sep;60(3):264-8. doi: 10.1016/j.annemergmed.2012.02.007. Epub 2012 Mar 15. PMID 22424652
- [Background] Bhisitkul DM, Listernick R, Shkolnik A, Donaldson JS, Henricks BD, Feinstein KA, Fernbach SK. Clinical application of ultrasonography in the diagnosis of intussusception. J Pediatr. 1992 Aug;121(2):182-6. doi: 10.1016/s0022-3476(05)81185-0. PMID 1640281
- [Background] Verschelden P, Filiatrault D, Garel L, Grignon A, Perreault G, Boisvert J, Dubois J. Intussusception in children: reliability of US in diagnosis--a prospective study. Radiology. 1992 Sep;184(3):741-4. doi: 10.1148/radiology.184.3.1509059.
- [Background] Williams H. Imaging and intussusception. Arch Dis Child Educ Pract Ed. 2008 Feb;93(1):30-6. doi: 10.1136/adc.2007.134304. No abstract available. PMID 18208983
- [Background] Ahn S, Park SH, Lee KH. How to demonstrate similarity by using noninferiority and equivalence statistical testing in radiology research. Radiology. 2013 May;267(2):328-38. doi: 10.1148/radiol.12120725. PMID 23610094